CLINICAL TRIAL: NCT04068259
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single Ascending Doses of PBI-4547 in Healthy Subjects
Brief Title: Single Ascending Dose Study of PBI-4547 in Healthy Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: PK data from first 3 cohorts does not support study continuation.There was no safety concerns
Sponsor: Liminal BioSciences Ltd. (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PBI-4547-CT-9-01; 180271 (Other: Syneos Health)
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — PBI-4547

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cohort 1, Dose 1 of PBI-4547 or Placebo (Experimental): Dose 1 of PBI-4547 or matching Placebo tablets by mouth
  Interventions: Drug: PBI-4547; Other: Placebo
- Cohort 2, Dose 2 of PBI-4547 or Placebo (Experimental): Dose 2 of PBI-4547 or matching Placebo tablets by mouth
  Interventions: Drug: PBI-4547; Other: Placebo
- Cohort 3, Dose 3 of PBI-4547 or Placebo (Experimental): Dose 3 of PBI-4547 or matching Placebo tablets by mouth
  Interventions: Drug: PBI-4547; Other: Placebo
- Cohort 4, Dose 4 of PBI-4547 or Placebo (Experimental): Dose 4 of PBI-4547 or matching Placebo tablets by mouth
  Interventions: Drug: PBI-4547; Other: Placebo
- Cohort 5, Dose 5 of PBI-4547 or Placebo (Experimental): Dose 5 of PBI-4547 or matching Placebo tablets by mouth
  Interventions: Drug: PBI-4547; Other: Placebo

INTERVENTIONS:
Drug: PBI-4547 — PBI-4547 tablet
Other: Placebo — Placebo tablet

SUMMARY:
This study will evaluate the safety, tolerability, and pharmacokinetics (PK) of PBI-4547 in healthy adult participants.

DETAILED DESCRIPTION:
This is a first-in-human, single-ascending dose study of PBI-4547 in healthy adult participants. PBI-4547 is a synthetic ligand of G protein-coupled receptor (GPR)40 and GPR84, which have been reported to play a role in fibrosis in various animal models as well as in tissue culture.

A total of 40 healthy adult participants will sequentially receive 1 of 5 doses of PBI-4547 (Dose1, 2, 3, 4 or 5) or matching placebo, with each cohort of 8 participants randomized in a 3:1 ratio to receive PBI-4547 or matching placebo.

A food-effect cohort will be added after review of the PK results of at least the first dose, and the following 2 doses, if needed. In this cohort participants will initially receive the study drug under fasting conditions (Period 1) followed by the same dose after the ingestion of a high-fat meal (Period 2) after a 14-day washout period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male participants or non-childbearing potential female participants, ≥18 and ≤55 years.
* Body mass index > 18.5 and < 30.0 kg/m^2, and body weight ≥ 50.0 kg for male participants and ≥ 45.0 kg for female participants.
* Continuous non-smoker who has not used tobacco or nicotine-containing products for at least 3 months prior to screening.
* Male participants with a pregnant partner must agree to use a condom from the first dosing until at least 90 days after study drug administration.
* Male participants must be willing not to donate sperm until 90 days after study drug administration.

Exclusion Criteria:

* Any clinically significant abnormality or abnormal laboratory test results.
* An estimated glomerular filtration rate (eGFR) <60 mL/min/1.73 m^2.
* Positive urine drug screen and history of significant drug abuse.
* History of significant allergic reactions to any drug.
* Use of any drugs known to induce or inhibit hepatic drug metabolism.
* Positive pregnancy test or breast-feeding participant.
* Clinically significant abnormalities in ECG, blood pressure, and heart rate at screening.
* History of significant alcohol abuse or regular use of alcohol.
* Use of medication other than topical products without significant systemic absorption.
* Donation of plasma.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-09-05 (Actual); Primary Completion 2019-10-08 (Actual); Study Completion 2019-10-08 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs) | 5-6 days
  TEAE is any untoward medical occurrence in a subject who has been administered a pharmaceutical product or not, which does not necessarily have a causal relationship with this treatment.
Number of participants with clinically significant laboratory evaluation findings | 5-6 days
  Laboratory tests for hematology, serum chemistry and urinalysis will be performed upon admission, at discharge, and at the follow-up visit (5 ± 1 day post-dose).
Number of participants with clinically significant electrocardiogram (ECG) Findings | 5-6 days
  Triplicate ECG will be performed upon admission, pre-dose, and approximately 1, 2, 8, and 24 hours post-dose, and at the follow-up visit (5 ± 1 day post-dose). Subjects will be continuously monitored using a Holter monitor from approximately 1 hour pre-dose until approximately 24 hours post-dose.
Number of participants with clinically significant vital sign findings | 5-6 days
  Vital signs include blood pressure, heart rate, respiratory rate, and oral body temperature will be measured upon admission, before discharge from the clinic and at the follow-up visit (5 ± 1 day post-dose).
Number of participants with physical examination findings | 5-6 days
  Brief physical examination will be conducted upon admission and at discharge. A complete physical examination will be conducted at screening and follow-up visit.

SECONDARY OUTCOMES:
AUC0-t for PBI-4547 | 48 hours
  Area under the concentration-time curve from time zero to the last non-zero concentration
AUC0-inf for PBI-4547 | 48 hours
  Area under the concentration-time curve from time zero to infinity (extrapolated)
Cmax for PBI-4547 | 48 hours
  Maximum observed concentration
Residual area for PBI-4547 | 48 hours
  Residual area calculated as 100*(1- AUC0-t / AUC0-inf)
Tmax for PBI-4547 | 48 hours
  Time of observed Cmax
T1/2 el for PBI-4547 | 48 hours
  Elimination half-life
Kel for PBI-4547 | 48 hours
  Elimination rate constant
Rkel for PBI-4547 | 48 hours
  Accumulation factor based on elimination rate constant
MRT for PBI-4547 | 48 hours
  Mean residence time
Cl/F for PBI-4547 | 48 hours
  Total body clearance, calculated as Dose/AUC0-inf;Cl/F normalized for subject body weight in kg will be calculated
Vd/F for PBI-4547 | 48 hours
  Apparent volume of distribution, calculated as Dose/(Kel x AUC0-inf). Vd/F normalized for subject body weight in kg will be calculated
AUC0-t for PBI-4547 under fed condition | 48 hours
  Area under the concentration-time curve from time zero to the last non-zero concentration after a high-fat diet
AUC0-inf for PBI-4547 under fed condition | 48 hours
  Area under the concentration-time curve from time zero to infinity (extrapolated) after a high-fat diet
Cmax for PBI-4547 under fed condition | 48 hours
  Maximum observed concentration after a high-fat diet
Tmax for PBI-4547 under fed condition | 48 hours
  Time of observed Cmax after a high-fat diet

CONTACTS AND LOCATIONS:
Overall Officials: John Moran, MD, Study Director — Prometic Pharma SMT Ltd.; Richard Larouche, MD, Principal Investigator — Syneos Health
Locations (2):
- Canada (2):
  - Syneos Health, Montreal, Quebec
  - Syneos Health, Québec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leduc M, Grouix B, Tremblay M, GervaisL, Sarra-Bournet F, Felton X, Simard J, Leblond FA, Laurin P and Gagnon L. PBI-4547 Improves Glucose Metabolism and Insulin Resistance, and Reduces Liver Damage in a High-Fat Diet Mouse Model of Obesity and Metabolic Syndrome. Diabetes 2018 Jul; 67(Supplement 1).
- [Background] Gagnon L, Laverdure A, Sarra-Bournet F, Cloutier M, Felton A, Treemblay M, Richard J, Gervais L, Laurin P, Leblond FA and Grouix B. PBI-4547 Reverses Diabetes and Metabolic Syndrome through Regulation of Lipid/Glucose Metabolism, ß-Oxidation and Fibrosis in Liver, and White Adipose Tissue in ob/ob Mice. Diabetes 2018 Jul; 67(Supplement 1).
- [Background] Sarra-Bournet F, Grouix B, Hince K, Felton A, Tremblay M, Abbott S, Duceppe JS, Zacharie B, Laurin P, Gagnon G. PBI-4547 decreases hepatic stellate cell activation via AMPK signaling pathway, and reduces fibrosis in carbon tetrachloride (CCL4)-induced hepatic fibrosis model. Journal of Hepatology 2018, 68:S365-S604.